CLINICAL TRIAL: NCT00621257
Title: Optimization of Vitamin D Stores and Its Impact on the Bone Health and Disease Outcomes of Children and Adolescents With IBD.
Brief Title: Vitamin D Levels in Children With IBD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Maintenance phase outcome unattenable
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Crohn's and Colitis Foundation (Other); NASPGHAN Foundation (Other Government)
Responsible Party: Principal Investigator, Helen Pappa, Assistant Professor, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1K23DK076979-01A1 (NIH); 1K23DK076979-01A1 (NIH)
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Results first posted 2017-02-17 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis
Keywords: IBD; Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis; Vitamin D
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Treatment A (Active Comparator): 2,000 IU/day of ergocalciferol orally for 6 weeks (control arm)
  Interventions: Dietary Supplement: ergocalciferol
- Treatment B (Experimental): 2,000 IU/day of cholecalciferol orally for 6 weeks
  Interventions: Dietary Supplement: Cholecalciferol
- Treatment C (Experimental): 50,000 IU of ergocalciferol once a week orally for 6 weeks
  Interventions: Dietary Supplement: ergocalciferol
- Maintenance A (Active Comparator): 400 IU/day of ergocalciferol orally over 2 years (control arm)
  Interventions: Dietary Supplement: ergocalciferol
- Maintenance B (Experimental): 2,000 IU/day of ergocalciferol orally from November 1 to April 30, and 1,000 IU/day of ergocalciferol orally for the remainder of the year over 2 years
  Interventions: Dietary Supplement: ergocalciferol

INTERVENTIONS:
Dietary Supplement: ergocalciferol — 8000 units/ml
  Other Names: Vitamin D2
  Arms: Maintenance A; Maintenance B; Treatment A; Treatment C
Dietary Supplement: Cholecalciferol — 400 units per drop
  Other Names: Vitamin D3
  Arms: Treatment B

SUMMARY:
Research has shown that children with Inflammatory Bowel Disease may have lower levels of vitamin D than healthy children, especially in the winter. Vitamin D is important for growing and maintaining healthy bones throughout life, and this is particularly important, since children with IBD frequently have low bone density. It may also be helpful in the treatment of IBD itself, because it helps reduce inflammation. Vitamin D levels are measured by the amount of 25 OHD in the blood; however, measuring this level on a regular basis is not yet the standard for children with IBD. The purpose of this study is to find the best way to treat low vitamin D levels, and to maintain good vitamin D levels throughout the year. It will also test whether having higher vitamin D levels will improve the bone health of children with IBD, and whether it will help them have milder disease.

DETAILED DESCRIPTION:
Vitamin D is essential for bone mineralization. The prevalence of vitamin D insufficiency [serum 25-hydroxy-vitamin D concentration (25OHD) ≤ 20 ng/mL] is high among adults with inflammatory bowel disease (IBD), and even higher in pediatric patients with IBD. Protein-losing enteropathy could represent both an etiologic factor for hypovitaminosis D, and an obstacle in treating it in IBD patients. There are currently no guidelines for the treatment of hypovitaminosis D in adults or children with IBD. Moreover we have obtained evidence that optimal vitamin D stores (25OHD ≥32 ng/mL) may not be maintained throughout the year in patients with IBD following current RDA recommendations. On the other hand, the prevalence of low bone mineral density is high among young patients with IBD, during a period in their lives when they should experience the most rapid acquisition of bone mass. Optimization of vitamin D status and its impact on the bone health of children with IBD has not been studied. In addition, vitamin D may play an important role in the regulation of the immune system as supported by animal models of colitis and in vitro human studies.

Prospective studies of the effect of vitamin D supplementation on disease outcomes have not been undertaken in children with IBD to date. We aim to perform a) a randomized controlled trial to compare the efficacy of 3 regimens in treating vitamin D insufficiency in pediatric patients with IBD over a period of 6 weeks. We will also evaluate the effects of each regimen on markers of bone resorption, bone formation and parathyroid hormone levels, and the relationship between the magnitude of gastrointestinal protein loss, as reflected by clearance of fecal alpha -1-antitrypsin, and the efficacy of the treatment. b) We also aim to perform a randomized controlled trial to compare the efficacy of 2 regimens of different doses of oral vitamin D2 in maintaining optimal vitamin D stores in pediatric patients with IBD over a period of 2 years. We intend to study the effect of each regimen on a) bone mass acquisition (measured via DXA and pQCT) and bone strength (measured via pQCT), b) bone formation and resorption markers and parathyroid hormone, and c) disease outcomes and disease severity over the same period of time.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of inflammatory bowel disease
* serum 25OHD level ≤ 20 ng/mL (Treatment Trial)
* serum 25OHD level > 20 ng/mL (Maintenance Trial)

Exclusion Criteria:

* Patients unable to take medications by mouth, pregnant, with liver/kidney failure, receiving anticonvulsant medications (specifically, phenobarbital, carbamazepine and phenytoin, since they lead to increased vitamin D metabolism through hepatic induction of the cytochrome P450 (CYP450) hydroxylase enzymes), regularly attending a tanning salon (once weekly or more), currently being treated for hypovitaminosis D with therapeutic doses of vitamin D (> 800 IU per day) and unwilling to discontinue this regimen.
* patients on growth hormone, anabolic steroid hormones, calcitonin, bisphosphonates (Maintenance Trial only)

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 134 (Actual)
Dates: Start 2008-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Pappa, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital, Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pappa HM, Mitchell PD, Jiang H, Kassiff S, Filip-Dhima R, DiFabio D, Quinn N, Lawton RC, Bronzwaer ME, Koenen M, Gordon CM. Maintenance of optimal vitamin D status in children and adolescents with inflammatory bowel disease: a randomized clinical trial comparing two regimens. J Clin Endocrinol Metab. 2014 Sep;99(9):3408-17. doi: 10.1210/jc.2013-4218. Epub 2014 Jun 13. PMID 24926949
- [Derived] Pappa HM, Mitchell PD, Jiang H, Kassiff S, Filip-Dhima R, DiFabio D, Quinn N, Lawton RC, Varvaris M, Van Straaten S, Gordon CM. Treatment of vitamin D insufficiency in children and adolescents with inflammatory bowel disease: a randomized clinical trial comparing three regimens. J Clin Endocrinol Metab. 2012 Jun;97(6):2134-42. doi: 10.1210/jc.2011-3182. Epub 2012 Mar 28. PMID 22456619

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment A: 2,000 IU/day of vitamin D2 orally for 6 weeks (control arm)
  ergocalciferol: 8000 units/ml
- Treatment B: 2,000 IU/day of vitamin D3 orally for 6 weeks
  Cholecalciferol: 400 units per drop
- Treatment C: 50,000 IU of vitamin D2 once a week orally for 6 weeks
  ergocalciferol: 8000 units/ml
- Maintenance A: 400 IU/day of vitamin D2 orally over 2 years (control arm)
  ergocalciferol: 8000 units/ml
- Maintenance B: 2,000 IU/day of vitamin D2 orally from November 1 to April 30, and 1,000 IU/day of vitamin D2 orally for the remainder of the year over 2 years
  ergocalciferol: 8000 units/ml
Period: Overall Study
Arm/Group | Treatment A | Treatment B | Treatment C | Maintenance A | Maintenance B
Started | 24 | 24 | 23 | 32 | 31
Completed | 20 | 21 | 20 | 26 | 22
Not Completed | 4 | 3 | 3 | 6 | 9
Not completed — Lost to Follow-up | 4 | 0 | 2 | 4 | 7
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A | Treatment B | Treatment C | Maintenance A | Maintenance B | Total
Number analyzed (Participants) | 24 | 24 | 23 | 32 | 31 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.9 (3) | 14.7 (3.5) | 16.3 (3.2) | 15.1 (3.1) | 14.5 (3.1) | 15.2 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 9 | 19 | 17 | 69
  Male | 14 | 10 | 14 | 13 | 14 | 65

OUTCOME MEASURES:

1. Primary Outcome: Treatment of Low 25 Hydroxy Vitamin D Levels in Pediatric Patients With Inflammatory Bowel Disease
Description: Change in serum 25OHD levels after treatment with vitamin D formulations for 6 weeks in pediatric patients with inflammatory bowel disease.
  25OHD is the most abundant vitamin D metabolite, which is bound to vitamin D binding protein. The measurement of its concentration in serum, reflects vitamin D stores.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 24 | 24 | 23
ng/ml | 9.3 (1.8) | 16.4 (2.0) | 25.4 (2.5)

2. Secondary Outcome: Maintenance of 25 Hydroxy Vitamin D Levels in Pediatric Patients With Inflammatory Bowel Disease
Description: Percentage of pediatric patients with inflammatory bowel disease who maintained their serum 25OHD level at or above 32 ng/mL at all study visits over the duration of the maintenance study 25OHD is the most abundant vitamin D metabolite, which is bound to vitamin D binding protein. The measurement of its concentration in serum, reflects vitamin D stores. Concentration at or above 32 ng/mL has been identified as optimal vitamin D level for bone health by majority of experts.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance A | Maintenance B
Number analyzed (Participants) | 32 | 31
Participants | 3 | 3

ADVERSE EVENTS:
Time Frame: 6 weeks while participant was on study medication for treatment trial
Description: For 1 year, while participant was on study medication for the maintenance trial.
Groups:
- Maintenance A: 400 IU per day of oral vitamin D2
  ergocalciferol 8000 IU/ml
- Maintenance B: 1,000 IU of oral vitamin D2 per day from May to October and 2,000 IU of oral vitamin D2 per day of oral vitamin D2 per day from November to April
  ergocalciferol 8000 IU/ml
Arm/Group | Treatment A | Treatment B | Treatment C | Maintenance A | Maintenance B
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/23 | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 5/24 | 8/24 | 4/23 | 19/32 | 15/31
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=24) | Treatment B (N=24) | Treatment C (N=23) | Maintenance A (N=32) | Maintenance B (N=31)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Drowsiness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 5 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Muscle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 3 (3)
headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 2 (2)
Increased thirst (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 5 (5)
Increased urination (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
itching skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
irregular heart beat (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss of appetite (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 4 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 5 (5) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
sensitive eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash on face and body (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Unusual tiredness, or weakness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Metallic taste (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Calcium deposit in tissues outside of bones (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes